CLINICAL TRIAL: NCT06957873
Title: Evaluation of the Relationship Between Craniovertebral Angle and Fibromyalgia Symptom Severity
Brief Title: Craniovertebral Angle and Fibromyalgia Severity
Status: Enrolling by invitation | Type: Observational
Sponsor: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Nadide Koca, Physical Medicine & Rehabilitation Specialist, Ankara Training and Research Hospital
Other Study IDs: AnkaraTRH-FTR-NK-06
Record Dates: First submitted 2025-04-27; First posted 2025-05-05 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-07

CONDITIONS: Craniovertebral Angle; Fibromyalgia Syndrome
Keywords: Fibromyalgia Syndrome; craniovertebral angle
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fibromyalgia Group: Fibromyalgia (FM) is a chronic pain syndrome characterized by widespread musculoskeletal pain, muscle stiffness, joint stiffness, insomnia, fatigue, mood disorders, cognitive dysfunction, anxiety, depression, and general sensitivity. Female and male patients between the ages of 18-55 who are diagnosed with FM according to the ACR 2010 diagnostic criteria will constitute the case group.
- Control Group: The control group, matching similar age and gender distribution, will be selected from patients presenting with mechanical knee pain complaints and without neck complaints. Considering the increased likelihood of degenerative changes in the cervical region with advancing age, the investigators limited the upper age limit to 55.

SUMMARY:
Forward Head Posture Frequency in Fibromyalgia Patients Assessed by Craniovertebral Angle: Association with Symptom Severity. Forward head posture is more common in patients with fibromyalgia and is a factor that increases symptom severity.

DETAILED DESCRIPTION:
Fibromyalgia (FM) is a chronic pain syndrome characterized by widespread musculoskeletal pain, muscle stiffness, joint rigidity, insomnia, fatigue, mood disorders, cognitive dysfunction, anxiety, depression, and general hypersensitivity.

Fibromyalgia is considered a central sensitivity syndrome. Central sensitization refers to a neuronal signal amplification mechanism within the central nervous system that leads to enhanced pain perception. Consequently, patients with FM exhibit an increased receptive field of pain, allodynia, and hyperalgesia.

Headache and temporomandibular disorders (TMD) are among the most common comorbidities in FM, displaying overlapping clinical and pathophysiological features.

Nociplastic pain is defined by the International Association for the Study of Pain as pain arising from altered nociception despite no clear evidence of actual or threatened tissue damage causing the activation of peripheral nociceptors or evidence for disease or lesion of the somatosensory system causing the pain. The mechanism of nociplastic pain is proposed to involve increased central nervous system sensitization and impaired sensory processing, accompanied by altered pain modulation. Definitive criteria for nociplastic pain have not yet been established. Eight specific disorders associated with central sensitization have been proposed: restless leg syndrome, chronic fatigue syndrome, FM, TMD, migraine or tension-type headache (TTH), irritable bowel syndrome, multiple chemical sensitivities, and whiplash injury.

Central sensitization is classically defined as a consequence of ongoing nociceptive inputs in chronic pain conditions. Its development is reported to be influenced by genetic factors, pain processing disorders in the brain, neuroendocrine and autonomic abnormalities, abnormal cytokines, and immune dysfunction.

As evident, conditions frequently accompanying FM, such as migraine, tension-type headache, chronic fatigue, irritable bowel syndrome, and TMD, share overlapping pathophysiology related to central sensitization.

A bidirectional relationship has been reported between primary headaches and craniocervical postural disorder, defined as Forward Head Posture (FHP). Postural disorders generate nociceptive peripheral stimuli that may lead to sensitization in the trigeminocervical complex.

The trigeminocervical complex (TCC), located in the brainstem, is a common convergence pathway where both trigeminal (dural) and cervical (primarily via the greater occipital nerve) afferent inputs are projected to higher centers in the thalamus and cortex. The TCC serves as the first sensory relay for meningeal and cephalic cutaneous information and forms the pathways for referred pain in primary headaches.

Brainstem interneurons have been shown to play a key role in pain modulation in migraine, TTH, and cluster headaches. Primary headache has been determined to result from trigeminocervical complex dysfunction. Neurophysiological studies on trigeminal reflexes support the concept of primary brainstem dysfunction and central hyperexcitability of trigeminal sensory pathways in chronic pain syndromes such as FM and TTH.

Similarly, animal studies in FM have identified a hyperalgesic state in the trigeminal region.

Sensitization in the trigeminocervical complex can lead to central sensitization by increasing thalamic and cortical stimulation. Peripheral and central sensitization are characterized by widespread hyperalgesia and allodynia. Consequently, patients with chronic primary headache exhibit a larger pain distribution area not only in the craniocervical region but throughout the entire spine.

The relationship between TCC sensitization and pain disorders has been well-documented in human and animal studies. Significant abnormalities in TCC responses have been observed in patients with trigeminal neuralgia, migraine, cluster headache, chronic tension-type headache, and fibromyalgia, attributed to hyperexcitability of trigeminal pathways.

Similarly, TMD, another comorbidity accompanying FM, frequently co-occurs with primary headaches, and the trigeminal system is reported to be the common pathophysiological mechanism.

Forward Head Posture (FHP) refers to the anterior displacement of the head relative to the trunk through upper cervical extension and lower cervical flexion. A craniovertebral angle (CVA) of 49° or less is defined as FHP.

FHP, characterized by forward head projection and rounded shoulders, is a common consequence of modern lifestyles involving prolonged use of laptops, mobile devices, or driving. It leads to persistent headache and is associated with migraine, TTH, and cervicogenic headaches.

The relationship between TMD and FHP is well-established. Forward head posture leads to TMD.

In the pathophysiology of primary headaches and TMD, which frequently accompany FM, the trigeminocervical complex emerges as a factor increasing central sensitization. FHP is reported to be a postural factor contributing to this. Central sensitization also plays a primary role in FM pathophysiology.

Postural studies in FM have reported increased thoracic kyphosis, lower CVA, and impaired cervical joint position sense.

To our knowledge, there are no studies examining the relationship between craniovertebral angle and disease severity in FM. We hypothesize that FHP may play a significant role in central sensitization in FM patients through the trigeminocervical complex, similar to its role in headaches and TMD. Therefore, we aim to investigate the frequency of FHP in FM patients and its relationship with FM disease severity.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-55 years
* Diagnosed with Fibromyalgia (FM) according to The American College of Rheumatology (ACR) 2010 Diagnostic Criteria for Fibromyalgia

Exclusion Criteria:

* History of past or current pathology in the cervical spine, thoracic spine, or upper extremities
* History of paraspinal or thoracic surgery involving the head, spine, or shoulders within the last six months
* Structural spinal malformation
* History of surgical or neurological disorders
* Cervical trauma or pain treatment within the last 6 months
* Temporomandibular surgery
* Psychiatric disorders (e.g., dementia, amnesia, or delirium)
* Systemic inflammatory rheumatic diseases

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Our research will be conducted as a prospective study. The case group will consist of male and female patients aged 18-55 years who present to the Physical Medicine and Rehabilitation clinic with widespread pain complaints and are diagnosed with Fibromyalgia (FM) according to ACR 2010 diagnostic criteria. The control group, matched for age and gender distribution, will be selected from patients presenting with mechanical knee pain complaints and no cervical symptoms. Considering the increased likelihood of degenerative changes in the cervical region with advancing age, the investigators limited the upper age limit to 55 years.
  Demographic data will be collected through face-to-face interviews during examination. During this time, patients will complete the Fibromyalgia Impact Questionnaire (FIQ). The FIQ is a 10-item questionnaire that evaluates the severity of fibromyalgia symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
The craniovertebral angle | up to 12 weeks
  During the same visit, permission will be obtained from patients for photography, and it will be explained that the photograph will be used solely for scientific research. One lateral photograph will be taken from consenting patients. For this purpose, the patient will be instructed to assume a standing posture and then relax. After the photographs taken with the camera placed at shoulder level are printed, the craniovertebral angle representing the forward head posture will be measured. The craniovertebral angle is the angle between the horizontal line passing through the 7th cervical vertebra and the line connecting the tragus of the ear to the C7 spinous process. The craniovertebral angle value will be calculated as the average value measured 5 times.

SECONDARY OUTCOMES:
Fibromyalgia Impact Questionnaire | up to 12 weeks
  The Fibromyalgia Impact Questionnaire (FIQ) consists of 10 items. The first item contains 11 questions related to physical function - each question is rated on a 4-point Likert-type scale. Items 2 and 3 ask the patient to mark the number of days they felt well and the number of days they could not work (including housework) due to fibromyalgia symptoms. Items 4 through 10 are horizontal linear scales marked in increments of 10 on which the patient rates work difficulty, pain, fatigue, morning tiredness, stiffness, anxiety, and depression. The highest possible score for each of the 10 items is 10, thus the highest possible score is 100. The average FM patient scores approximately 50 points; severely affected patients typically score ≥70 points.

CONTACTS AND LOCATIONS:
Overall Officials: Nadide Koca, M.D., Principal Investigator — Ankara Training and Research Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Department of Physical Therapy and Rehabilitation, University of Health Sciences, Ankara Training and Research Hospital, Ankara, Altindag
  - University of Health Sciences, Ankara Training and Research Hospital, Ankara, Altindag

REFERENCES:
- [Background] Graff-Radford SB, Abbott JJ. Temporomandibular Disorders and Headache. Oral Maxillofac Surg Clin North Am. 2016 Aug;28(3):335-49. doi: 10.1016/j.coms.2016.03.004. PMID 27475510
- [Background] Abanoz Y, Gulen Abanoz Y, Gunduz A, Karadeniz D, Erdemir Kiziltan M. Long latency trigemino-cervical reflex in restless legs syndrome. Int J Neurosci. 2024 Aug;134(8):924-930. doi: 10.1080/00207454.2022.2158826. Epub 2022 Dec 28. PMID 36533413
- [Background] Deodato M, Granato A, Del Frate J, Martini M, Manganotti P. Differences in musculoskeletal dysfunctions and in postural alterations between chronic migraine and chronic tension type headache: A cross-sectional study. J Bodyw Mov Ther. 2024 Jan;37:404-411. doi: 10.1016/j.jbmt.2023.11.011. Epub 2023 Nov 17. PMID 38432837
- [Background] Nazeri M, Zarei MR, Pourzare AR, Ghahreh-Chahi HR, Abareghi F, Shabani M. Evidence of Altered Trigeminal Nociception in an Animal Model of Fibromyalgia. Pain Med. 2018 Feb 1;19(2):328-335. doi: 10.1093/pm/pnx114. PMID 28505350
- [Background] Wodehouse T, Bahra A, Mehta V. Changes in peripheral and central sensitization in patients undergoing occipital nerve stimulation. Br J Pain. 2020 Nov;14(4):250-255. doi: 10.1177/2049463719860548. Epub 2019 Jul 29. PMID 33194189
- [Background] Caponnetto V, Deodato M, Robotti M, Koutsokera M, Pozzilli V, Galati C, Nocera G, De Matteis E, De Vanna G, Fellini E, Halili G, Martinelli D, Nalli G, Serratore S, Tramacere I, Martelletti P, Raggi A; European Headache Federation School of Advanced Studies (EHF-SAS). Comorbidities of primary headache disorders: a literature review with meta-analysis. J Headache Pain. 2021 Jul 14;22(1):71. doi: 10.1186/s10194-021-01281-z. PMID 34261435
- [Background] Liang Z, Galea O, Thomas L, Jull G, Treleaven J. Cervical musculoskeletal impairments in migraine and tension type headache: A systematic review and meta-analysis. Musculoskelet Sci Pract. 2019 Jul;42:67-83. doi: 10.1016/j.msksp.2019.04.007. Epub 2019 Apr 25. PMID 31054485
- [Background] Ji RR, Nackley A, Huh Y, Terrando N, Maixner W. Neuroinflammation and Central Sensitization in Chronic and Widespread Pain. Anesthesiology. 2018 Aug;129(2):343-366. doi: 10.1097/ALN.0000000000002130. PMID 29462012
- [Background] Yoo YM, Kim KH. Current understanding of nociplastic pain. Korean J Pain. 2024 Apr 1;37(2):107-118. doi: 10.3344/kjp.23326. Epub 2024 Mar 20. PMID 38504389
- [Background] Yakkaphan P, Smith JG, Chana P, Tan HL, Ravindranath PT, Lambru G, Renton T. Temporomandibular Disorders and Fibromyalgia Prevalence: A Systematic Review and Meta-Analysis. J Oral Facial Pain Headache. 2023 Nov 17;37(3):177-193. doi: 10.11607/ofph.3260. PMID 37975782
- [Background] Lee W, Shin HJ, Min IK, Kim CS, Kim KM, Heo K, Chu MK. Shared comorbidity of depression, migraine, insomnia, and fibromyalgia in a population-based sample. J Affect Disord. 2024 Jun 1;354:619-626. doi: 10.1016/j.jad.2024.03.077. Epub 2024 Mar 15. PMID 38494140
- [Background] Siracusa R, Paola RD, Cuzzocrea S, Impellizzeri D. Fibromyalgia: Pathogenesis, Mechanisms, Diagnosis and Treatment Options Update. Int J Mol Sci. 2021 Apr 9;22(8):3891. doi: 10.3390/ijms22083891. PMID 33918736
- [Background] de Tommaso M, Vecchio E, Nolano M. The puzzle of fibromyalgia between central sensitization syndrome and small fiber neuropathy: a narrative review on neurophysiological and morphological evidence. Neurol Sci. 2022 Mar;43(3):1667-1684. doi: 10.1007/s10072-021-05806-x. Epub 2022 Jan 14. PMID 35028777
- [Background] Oton T, Carmona L, Rivera J. Patient-journey of fibromyalgia patients: A scoping review. Reumatol Clin (Engl Ed). 2024 Feb;20(2):96-103. doi: 10.1016/j.reumae.2023.07.005. PMID 38395498